CLINICAL TRIAL: NCT03610048
Title: A Phase 3b Extension Study of Adjunctive ALKS 5461 in the Treatment of Refractory Major Depressive Disorder
Brief Title: A Long Term Study of ALKS 5461 in the Treatment of Refractory Major Depressive Disorder (MDD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALK5461-218
Record Dates: First submitted 2018-07-26; First posted 2018-08-01 (Actual); Results first posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-06

CONDITIONS: Refractory Major Depressive Disorder
Keywords: Alkermes; Major depressive disorder; Depression; ALKS 5461
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — ALKS 5461

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALKS 5461 (Experimental): Sublingual tablets
  Interventions: Drug: ALKS 5461

INTERVENTIONS:
Drug: ALKS 5461 — samidorphan + buprenorphine administered sublingually

SUMMARY:
This study will assess the long-term safety and tolerability of ALKS 5461 as an adjunctive treatment for refractory MDD.

ELIGIBILITY:
Inclusion Criteria:

* Completed study ALK5461-217
* Be willing to abide by the contraception requirements as outlined in the study protocol
* Be willing and able to follow the study procedures and visits as outlined in the protocol
* Additional criteria may apply

Exclusion Criteria:

* Pregnant, planning to become pregnant, or breastfeeding
* A positive urine drug test for drugs of abuse
* Poses a current suicide risk
* Additional criteria may apply

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkermes Medical Director, Study Director — Alkermes, Inc.
Locations (33):
- United States (29):
  - Alkermes Investigational Site, Tucson, Arizona
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Los Alamitos, California
  - Alkermes Investigational Site, Oceanside, California
  - Alkermes Investigational Site, Pico Rivera, California
  - Alkermes Investigational Site, Redlands, California
  - Alkermes Investigational Site, Santa Ana, California
  - Alkermes Investigational Site, Sherman Oaks, California
  - Alkermes Investigational Site, Temecula, California
  - Alkermes Investigational Site, Hollywood, Florida
  - Alkermes Investigational Site, Jacksonville, Florida
  - Alkermes Investigational Site, Lauderhill, Florida
  - Alkermes Investigational Site, Orlando, Florida
  - Alkermes Investigational Site, Palm Bay, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Decatur, Georgia
  - Alkermes Investigational Site, Pikesville, Maryland
  - Alkermes Investigational Site, O'Fallon, Missouri
  - Alkermes Investigational Site, Jamaica, New York
  - Alkermes Investigational Site, Mount Kisco, New York
  - Alkermes Investigational Site, Canton, Ohio
  - Alkermes Investigational Site, Cincinnati, Ohio
  - Alkermes Investigational Site, Oklahoma City, Oklahoma
  - Alkermes Investigational Site, Allentown, Pennsylvania
  - Alkermes Investigational Site, Memphis, Tennessee
  - Alkermes Investigational Site, Dallas, Texas
  - Alkermes Investigational Site, DeSoto, Texas
  - Alkermes Investigational Site, Woodstock, Vermont
  - Alkermes Investigational Site, Bellevue, Washington
- Australia (3):
  - Alkermes Investigational Site, Frankston, Victoria
  - Alkermes Investigational Site, Noble Park, Victoria
  - Alkermes Investigational Site, Richmond, Victoria
- Alkermes Investigational Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects that had completed the 12-week treatment period in the antecedent study ALK5461-217 were eligible to be enrolled in the study.
Pre-assignment Details: A total of 175 patients were administered at least one dose of ALKS 5461 and included in the safety population.
Groups:
- ALKS 5461: All subjects assigned to ALKS 5461
  Sublingual tablets
  ALKS 5461: samidorphan + buprenorphine administered sublingually
Period: Overall Study
Arm/Group | ALKS 5461
Started | 175
Completed Treatment | 15
Completed (Completed study) | 14
Not Completed | 161
Not completed — Study terminated by sponsor | 84
Not completed — Adverse Event | 32
Not completed — Withdrawal by Subject | 31
Not completed — Lost to Follow-up | 8
Not completed — Other | 4
Not completed — Physician Decision | 1
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Arm/Group | ALKS 5461
Number analyzed (Participants) | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (12.87)
Age, Customized [Count of Participants; unit: Participants]
  <55 years | 127
  >=55 years | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122
  Male | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 151
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 148
  More than one race | 3
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 142
  Australia | 23
  Puerto Rico | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs)
Description: Number and percentage of subjects experiencing TEAEs
Time Frame: Up to 68 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ALKS 5461
Number analyzed (Participants) | 175
Participants | 108

ADVERSE EVENTS:
Time Frame: 90 weeks
Arm/Group | ALKS 5461
All-Cause Mortality (participants affected / at risk) | 0/175
Serious Adverse Events (participants affected / at risk) | 4/175
Other Adverse Events (participants affected / at risk) | 85/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALKS 5461 (N=175)
Vomiting (Gastrointestinal disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALKS 5461 (N=175)
Nausea (Gastrointestinal disorders) | 36
Constipation (Gastrointestinal disorders) | 17
Vomiting (Gastrointestinal disorders) | 16
Dry mouth (Gastrointestinal disorders) | 8
Abdominal pain upper (Gastrointestinal disorders) | 4
Dizziness (Nervous system disorders) | 21
Headache (Nervous system disorders) | 12
Sedation (Nervous system disorders) | 12
Somnolence (Nervous system disorders) | 9
Dysgeusia (Nervous system disorders) | 6
Upper respiratory tract infection (Infections and infestations) | 10
Urinary tract infection (Infections and infestations) | 7
Nasopharyngitis (Infections and infestations) | 5
Insomnia (Psychiatric disorders) | 7
Fatigue (General disorders) | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6
Vertigo (Ear and labyrinth disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT03610048/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT03610048/SAP_001.pdf